CLINICAL TRIAL: NCT02996591
Title: Spinal Versus General Anesthesia With Popliteal and Adductor Canal Blocks for Ambulatory Foot and Ankle Surgery: A Double-Blinded Randomized Controlled Trial.
Brief Title: Spinal Versus General Anesthesia With Popliteal and Adductor Canal Blocks for Ambulatory Foot and Ankle Surgery.
Acronym: LMA vs Spinal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-0499
Record Dates: First submitted 2016-12-02; First posted 2016-12-19 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Nerve Block; General Anesthesia; Spinal Anesthesia; Pain; Postoperative Nausea and Vomiting
Keywords: Nerve Block; General Anesthesia; Spinal Anesthesia; Pain; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Pain; Postoperative Nausea and Vomiting | interventions — Bupivacaine; Dexamethasone; Midazolam; Glycopyrrolate; Ketamine; Propofol; Health Services Needs and Demand; Mepivacaine; Anesthesia, Spinal; Sevoflurane; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Spinal anesthesia with popliteal and adductor canal blocks. (Active Comparator): Ultrasound (US) guided sciatic nerve blocks in the popliteal fossa and adductor canal block with 25 mL and 10 mL, respectively, of 0.25% bupivacaine (plus 2 mg preservative-free (PF) dexamethasone / 30 ml), performed under procedural IV sedation protocol. IV sedation protocol: midazolam, 2-5 mg IV + Glycopyrrolate, 0.1 mg IV + Ketamine, 10-20 mg, + propofol as needed. Spinal protocol: 45-60 mg 1.5% mepivacaine, depending on the expected case duration (45 mg for cases with projected duration 1-2 hours, 60 mg for cases with projected duration 2-3 hours). Intraoperative sedation maintained with propofol infusion and ketamine, 10 mg/hr.
  Interventions: Procedure: 25 mL of 0.25% bupivacaine plus 2 mg preservative-free (PF) dexamethasone / 30 ml for popliteal nerve block; Procedure: 10 mL of 0.25% bupivacaine plus 2 mg preservative-free (PF) dexamethasone / 30 ml for adductor canal nerve block; Drug: Midazolam, 2-5 mg IV + Glycopyrrolate, 0.1 mg IV + Ketamine, 10-20 mg + propofol as needed; Procedure: 45-60 mg of 1.5% mepivacaine for spinal anesthesia
- General anesthesia with popliteal and adductor canal blocks. (Active Comparator): Ultrasound (US) guided sciatic nerve blocks in the popliteal fossa and adductor canal block with 25 mL and 10 mL, respectively, of 0.25% bupivacaine (plus 2 mg preservative-free (PF) dexamethasone / 30 ml), performed under procedural IV sedation protocol. IV sedation protocol: midazolam, 2-5 mg IV + Glycopyrrolate, 0.1 mg IV + Ketamine, 10-20 mg, + propofol as needed. General anesthesia protocol: After induction with propofol and insertion of the LMA, anesthesia maintained with titrated propofol infusion, sevoflurane, ketamine 10 mg/hr.
  Interventions: Procedure: 25 mL of 0.25% bupivacaine plus 2 mg preservative-free (PF) dexamethasone / 30 ml for popliteal nerve block; Procedure: 10 mL of 0.25% bupivacaine plus 2 mg preservative-free (PF) dexamethasone / 30 ml for adductor canal nerve block; Drug: Midazolam, 2-5 mg IV + Glycopyrrolate, 0.1 mg IV + Ketamine, 10-20 mg + propofol as needed; Procedure: LMA insertion + titrated propofol infusion + sevoflurane + ketamine 10 mg/hr for general anesthesia

INTERVENTIONS:
Procedure: 25 mL of 0.25% bupivacaine plus 2 mg preservative-free (PF) dexamethasone / 30 ml for popliteal nerve block
Procedure: 10 mL of 0.25% bupivacaine plus 2 mg preservative-free (PF) dexamethasone / 30 ml for adductor canal nerve block
Drug: Midazolam, 2-5 mg IV + Glycopyrrolate, 0.1 mg IV + Ketamine, 10-20 mg + propofol as needed
Procedure: 45-60 mg of 1.5% mepivacaine for spinal anesthesia
  Arms: Spinal anesthesia with popliteal and adductor canal blocks.
Procedure: LMA insertion + titrated propofol infusion + sevoflurane + ketamine 10 mg/hr for general anesthesia
  Arms: General anesthesia with popliteal and adductor canal blocks.

SUMMARY:
The purpose of this study is to determine if there is a difference in patient outcomes with general anesthesia versus spinal anesthesia when given in addition to popliteal and adductor canal nerve blocks for foot and ankle surgery. Popliteal and adductor canal nerve blocks are injections of local anesthetic agents near nerves in the back and front of the knee going to the foot and ankle that provide numbness during and after surgery. These peripheral nerve blocks offer good pain control and reduce the need for opioids (opioids are pain medications such as morphine, Dilaudid, and oxycodone). General anesthesia involves the flow of oxygen and anesthesia gas through a tube which, along with additional intravenous medications, causes unconsciousness and unawareness of sensations during surgery. Spinal anesthesia involves an injection of local anesthetic in the lower back, which causes numbness below the waist. In addition to spinal anesthesia, a sedative is typically given intravenously to cause relaxation and sleepiness throughout surgery.

General, spinal, and nerve block anesthesia are all routinely used for surgery at the Hospital for Special Surgery. General or spinal anesthesia is typically used in addition to peripheral nerve blocks during foot and ankle surgery to 1) allow the surgeons to use a thigh tourniquet to reduce bleeding, 2) provide anesthesia earlier, and 3) prevent unwanted movement. However, it is unclear whether general or spinal anesthesia provides better patient outcomes when given with peripheral nerve blocks. Some reports show that on its own, spinal anesthesia has advantages over general anesthesia in terms of side effects such as nausea and pain. However, these advantages may also be gained from combining peripheral nerve blocks with general anesthesia. Spinal anesthesia can be associated with headache and backache, although headache and backache can also happen after operations performed with general anesthesia. A previous study at the Hospital for Special Surgery showed low rates of nausea among patients who received nerve blocks with spinal anesthesia, and no nausea among patients who received a nerve block with general anesthesia. Therefore, the primary aim of this study is to determine if, as a treatment, either general or spinal anesthesia has advantages over the other treatment in terms of readiness for discharge, side effects, pain and patient satisfaction in an ambulatory foot and ankle population.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 aged patients
* American Society of Anesthesiologists (ASA) Physical Status classification 1-3
* Elective foot and ankle day surgery procedures, lasting between 1 and 3 hours as per surgeon, performed by 3 co-investigator surgeons.
* Planned for combined popliteal and adductor canal block
* No contraindications for spinal or LMA general anesthesia

Exclusion Criteria:

* Incapable of providing informed consent
* Contraindications for regional or LMA anesthesia (anticoagulation, infection at injection site)
* Anticipated difficult airway
* BMI>40
* Anticipated surgical procedure time less than 1 hour or more than 3 hours
* Hx of severe postoperative nausea and vomiting
* ASA >3
* Peripheral neuropathy affecting the operative extremity
* Pregnant or nursing women
* Chronic opioid use (daily use of opioids one month prior to surgery/ patients requiring chronic pain interventions)
* Prone position
* Obstructive sleep apnea with planned admission overnight to the hospital
* Known allergy/sensitivity to any study medications
* Planned admission after surgery
* Non-English speaking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques YaDeau, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, New York, United States

REFERENCES:
- [Derived] YaDeau JT, Fields KG, Kahn RL, LaSala VR, Ellis SJ, Levine DS, Paroli L, Luu TH, Roberts MM. Readiness for Discharge After Foot and Ankle Surgery Using Peripheral Nerve Blocks: A Randomized Controlled Trial Comparing Spinal and General Anesthesia as Supplements to Nerve Blocks. Anesth Analg. 2018 Sep;127(3):759-766. doi: 10.1213/ANE.0000000000003456. PMID 29847387

RESULTS

PARTICIPANT FLOW:
Groups:
- Spinal Anesthesia With Popliteal and Adductor Canal Blocks.: Ultrasound (US) guided sciatic nerve blocks in the popliteal fossa and adductor canal block with 25 mL and 10 mL, respectively, of 0.25% bupivacaine (plus 2 mg preservative-free (PF) dexamethasone / 30 ml), performed under procedural IV sedation protocol: midazolam, 2-5 mg IV + Glycopyrrolate, 0.1 mg IV + Ketamine, 10-20 mg, + propofol as needed. Spinal protocol: 45-60 mg 1.5% mepivacaine, depending on the expected case duration (45 mg for cases with projected duration 1-2 hours, 60 mg for cases with projected duration 2-3 hours). Intraoperative sedation maintained with propofol infusion and ketamine, 10 mg/hr.
  25 mL of 0.25% bupivacaine plus 2 mg preservative-free (PF) dexamethasone / 30 ml for popliteal nerve block
  10 mL of 0.25% bupivacaine plus 2 mg preservative-free (PF) dexamethasone / 30 ml for adductor canal nerve block
  Midazolam, 2-5 mg IV + Glycopyrrolate, 0.1 mg IV + Ketamine, 10-20 mg + propofol as needed
  45-60 mg of 1.5% mepivacaine for
- General Anesthesia With Popliteal and Adductor Canal Blocks.: Ultrasound (US) guided sciatic nerve blocks in the popliteal fossa and adductor canal block with 25 mL and 10 mL, respectively, of 0.25% bupivacaine (plus 2 mg preservative-free (PF) dexamethasone / 30 ml), performed under procedural IV sedation protocol. IV sedation protocol: midazolam, 2-5 mg IV + Glycopyrrolate, 0.1 mg IV + Ketamine, 10-20 mg, + propofol as needed. General anesthesia protocol: After induction with propofol and insertion of the LMA, anesthesia maintained with titrated propofol infusion, sevoflurane, ketamine 10 mg/hr.
  25 mL of 0.25% bupivacaine plus 2 mg preservative-free (PF) dexamethasone / 30 ml for popliteal nerve block
  10 mL of 0.25% bupivacaine plus 2 mg preservative-free (PF) dexamethasone / 30 ml for adductor canal nerve block
  Midazolam, 2-5 mg IV + Glycopyrrolate, 0.1 mg IV + Ketamine, 10-20 mg + propofol as needed
  LMA insertion + titrated propofol infusion + sevoflurane + ketamine 10 mg/hr for general anesthesia
Period: Overall Study
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks. | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 18 | 32
  >=65 years | 4 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (13) | 47 (11) | 51 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 16 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Time Until Patient is Ready for Discharge From Post-Anesthesia Care Unit (PACU) to Home.
Description: Modified Aldrete Scoring System and Marshall and Chung Postanesthesia Discharge Scoring System, measured in time until discharge criteria is met (in minutes)
Time Frame: Duration of stay in recovery room after surgery
Measure: Mean (Inter-Quartile Range); unit: Minutes
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 18
Minutes | 81 [55 to 104] | 43.5 [38 to 71]

2. Secondary Outcome: Numerical Rating Scale (NRS) Pain Scores at 1 Hour Postop
Description: NRS Pain scores at 1 hour after surgery. Rated on a scale of 0 (no pain) to 10 (worst pain imaginable).
Time Frame: 1 hour after PACU admission
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 18
units on a scale | 0 (0) | 1.8 (2.1)

3. Secondary Outcome: Numerical Rating Scale Pain Scores at 2 Hours Postop
Description: Numerical rating scale pain score as reported by the patient at 2 hours post-operatively. Rated on a scale of 0 (no pain) to 10 (worst pain imaginable).
Time Frame: 2 hours after PACU admission
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 18
units on a scale | .4 (1.3) | .9 (1.6)

4. Secondary Outcome: Numerical Rating Scale Pain Scores on Postoperative Day (POD) 1
Description: Numerical Rating Scale Pain from 0-10. 0 being no pain at all. 10 being the worst pain imaginable.
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 17
score on a scale | 1 (1.6) | 1 (1.7)

5. Secondary Outcome: Postoperative Discomfort and Needs (Post-op Pain, Sore Throat, Back Pain, Nausea, Cold, Hunger, Thirst)
Description: Leiden Perioperative Care Patient Satisfaction questionnaire (LPPSq) score. Performed at 1 hour postoperatively. To what degree did patients have the following symptoms. Rated 1-5, 1 being not at all. 5 being extremely.
Time Frame: 1 hour after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 17
score on a scale
  Pain | 1.1 (.5) | 1.6 (.8)
  A Sore Throat | 1.2 (.5) | 1.6 (1.1)
  Back Pain | 1.2 (.5) | 1.2 (.5)
  Vomiting | 1 (0) | 1 (0)
  Cold | 1.4 (.8) | 1.3 (.6)
  Hunger | 1.9 (1.2) | 1.7 (.9)
  Thirst | 2.7 (1.2) | 2.5 (1.2)

6. Secondary Outcome: Postoperative Discomfort and Needs (Post-op Pain, Sore Throat, Back Pain, Nausea, Cold, Hunger, Thirst)
Description: Rating the Nausea/Vomiting of patients post-operatively.
Time Frame: 2 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 18
score on a scale
  Pain | 1.2 (.5) | 1.4 (.7)
  Sore Throat | 1.2 (.4) | 1.6 (1.1)
  Back Pain | 1.1 (.2) | 1.2 (.5)
  Vomiting | 1 (0) | 1 (0)
  Cold | 1.1 (.3) | 1.1 (.2)
  Hunger | 1.4 (.7) | 1.2 (.5)
  Thirst | 2.1 (1.2) | 1.8 (1.2)

7. Secondary Outcome: Postoperative Discomfort and Needs (Post-op Pain, Sore Throat, Back Pain, Nausea, Cold, Hunger, Thirst)
Description: Leiden Perioperative Care Patient Satisfaction questionnaire (LPPSq). From 1-5. 1 being not at all. 5 being extremely.
Time Frame: Postoperative day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 17
score on a scale
  Pain | 1.4 (.7) | 1.5 (.6)
  Sore Throat | 1.2 (.4) | 1.5 (.6)
  Back Pain | 1.1 (.3) | 1.2 (.6)
  Vomiting | 1 (0) | 1 (0)
  Cold | 1.3 (.6) | 1 (0)
  Hunger | 1.4 (.7) | 1.7 (.7)
  Thirst | 2.3 (1) | 2.2 (1)

8. Secondary Outcome: Incidence of Post-dural Puncture Headache
Time Frame: Postoperative day 1 and if present, monitored until resolution
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 17
Participants
  Yes | 4 | 3
  No | 14 | 14

9. Secondary Outcome: Incidence of Transient Neurologic Symptoms
Time Frame: Postoperative day 1 and if present, monitored until resolution
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 18
Participants
  Normal | 18 | 18
  Transient Neurological Symptoms | 0 | 0

10. Secondary Outcome: Opioid Consumption
Description: Opioid consumption (mg OME) during inpatient stay
Time Frame: Duration of stay in recovery room after surgery (average 2 hours)
Measure: Mean (Standard Deviation); unit: mg OME
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 18
mg OME | 2.2 (7.3) | 5 (7)

11. Secondary Outcome: Opioid Consumption Through First Postoperative Day. Measured in mg OME
Time Frame: Postoperative day 1
Measure: Mean (Standard Deviation); unit: mg OME
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 17
mg OME | 8.3 (10.3) | 11 (12.3)

12. Secondary Outcome: Non-opioid Analgesic Consumption
Description: The number of patients who took non-opioid analgesic medication for post-operative pain between hospital discharge and postoperative day 1.
Time Frame: Hospital discharge to postoperative day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 17
Participants
  yes | 12 | 12
  No | 6 | 5

13. Secondary Outcome: Opioid-Related Symptom Distress Scale (ORSDS) Score
Description: Opioid-related symptom distress scale. The ORSDS measures patient opioid-related symptoms on a 4-point scale that evaluates 3 symptom distress dimension (severity, frequency, and bothersomeness) for 12 opioid-related symptoms. Scores range from 0-4, and the mean of the 12 answers is the ORSDS score. Higher values indicate worse opioid-related symptoms.
Time Frame: 2 hours after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 17
units on a scale | .3 (.2) | .3 (.3)

14. Secondary Outcome: Cognitive Recovery
Description: Postoperative Quality Recovery Scale Cognitive Domain questionnaire. Asked at 1 hour post-operatively. Either yes (return to pre-operative cognitive function levels) or no (not yet returned to pre-operative function levels)
Time Frame: 1 hour after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 17 | 17
Participants
  No | 3 | 4
  Yes | 14 | 13

15. Secondary Outcome: Incidence of Urinary Catheterization
Time Frame: Duration of stay in recovery room after surgery (average 2 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 18
Participants
  Yes | 0 | 0
  No | 18 | 18

16. Secondary Outcome: Anesthesia-related Postoperative Complications
Description: Measuring any anesthesia-related post-op complications that occured (yes or no)
Time Frame: Surgery start to postoperative day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 18
Participants
  Yes | 0 | 0
  No | 18 | 18

17. Secondary Outcome: Assessment of Patient Blinding to Group Assignment
Description: Patients will be asked whether they believe they were in the general anesthesia or spinal anesthesia group. These responses are then validated using the Bang Blinding Index, which either confirms or refutes the validity of the blinding. The scale runs from -1 to 1, with a score of 0 indicating complete blinding, -1 indicating opposite guessing of groups, and 1 indicating a complete lack of blinding.
Time Frame: Postoperative day 1
Measure: Number (95% Confidence Interval); unit: Bang blinding index
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 17
Bang blinding index | .588 [.313 to .864] | .722 [.47 to .974]
Statistical Analysis 1: Comparison: Spinal Anesthesia With Popliteal and Adductor Canal Blocks. vs General Anesthesia With Popliteal and Adductor Canal Blocks; Test type: Other; p = .038, Regression, Logistic; generalized estimating equations method = 45
Statistical Analysis 2: Comparison: Spinal Anesthesia With Popliteal and Adductor Canal Blocks. vs General Anesthesia With Popliteal and Adductor Canal Blocks; Test type: Other — Bang blinding index; p < .001, Bang Blinding Index; 95% confidence interval

18. Secondary Outcome: Patient Satisfaction
Description: Yes/no if patients would request the same anesthetic that they received
Time Frame: POD1
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 17
Participants
  Yes | 18 | 17
  No | 0 | 0

19. Secondary Outcome: Cognitive Recovery at 2 Hours Post-operative
Description: Postoperative Quality Recovery Scale Cognitive Domain questionnaire. Asked at 2 hour post-operatively. Either yes (return to pre-operative cognitive function levels) or no (not yet returned to pre-operative function levels)
Time Frame: 2 hours after PACU admission
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 17 | 17
Participants
  No | 1 | 4
  Yes | 16 | 13

20. Secondary Outcome: Cognitive Recovery on POD1
Description: Postoperative Quality Recovery Scale Cognitive Domain questionnaire. Asked on postoperative day 1. Either yes (return to pre-operative cognitive function levels) or no (not yet returned to pre-operative function levels)
Time Frame: Postoperative day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 17 | 17
Participants
  No | 3 | 2
  Yes | 14 | 15

21. Secondary Outcome: Nausea Intensity
Description: Nausea intensity ranked on NRS score following PACU admission to 2 hours after discharge. Scored from 0-10. 0 Being no nausea, 10 being worst nausea imaginable.
Time Frame: 2 hours after PACU admission
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 18
score on a scale | 0 [0 to 0] | 0 [0 to 0]

22. Secondary Outcome: Back Pain on POD1
Description: Back pain (yes/no) on POD1
Time Frame: Postoperative day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
Number analyzed (Participants) | 18 | 17
Participants
  No | 16 | 14
  Yes | 2 | 3

ADVERSE EVENTS:
Time Frame: 24 hours postoperatively.
Description: Does not differ
Arm/Group | Spinal Anesthesia With Popliteal and Adductor Canal Blocks. | General Anesthesia With Popliteal and Adductor Canal Blocks.
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT02996591/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT02996591/Prot_SAP_001.pdf